CLINICAL TRIAL: NCT03990129
Title: Single-center, Open, Controlled Study to Investigate the Interaction of Metamizole With the Cytochrome p450 System in Healthy Subjects by Application of the Basel Cocktail
Brief Title: Pharmacokinetic Interactions of Metamizole (Dipyrone) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-00753
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Inhibition; Induction; Drug-Drug Interaction
Keywords: Metamizole; Dipyrone; Basel Cocktail; Drug-Drug Interaction; Phenotyping
MeSH Terms: conditions — Inhibition, Psychological | interventions — Dipyrone

STUDY DESIGN:
Intervention Model Description: Two phase study, before-after comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study population (Other): All participants
  Interventions: Drug: Metamizole

INTERVENTIONS:
Drug: Metamizole — One week treatment with metamizole (500 mg tablets, 2-2-2)

SUMMARY:
Investigators conducted a single center, two-phased, open, controlled pharmacokinetic study to investigate the drug-drug interaction potential of metamizole. For this reason, healthy male volunteers were screened.

Enrolled participants were phenotyped on day 1 using the Basel Cocktail (phenotyping cocktail containing specific substrates for CYP1A2, CYP2B6, CYP2C9, CYP2C19, CYP2D6, CYP3A4). After, they received metamizole treatment for 8 days (3 grams per day). On the 8th day (day 9), they were phenotyped again with the Basel Cocktail and the respective phenotypes (d1 vs. d9) were compared.

DETAILED DESCRIPTION:
12 healthy male subjects meeting the inclusion and exclusion criteria were enrolled. On day 1, they ingested a capsule containing the Basel Cocktail (1A2: caffeine, 2B6: efavirenz, 2C9: flurbiprofen, 2C19: omeprazole, 2D6: metoprolol, 3A4: midazolam) in fastened state. Blood samples were withdrawn over 24 hours and the AUC ratios between metabolite and parent were calculated to determine the phenotype.

Probands began metamizole treatment (3000 mg/day) at the day of the 24h measurement. After 3-4 day, probands were returning to the facility to ensure safety during the metamizole treatment, blood cell count and metamizole metabolites were measured. After the 7 days of treatment, probands were exposed again to the Basel Cocktail in a fastened state. Probands were still exposed to metamizole to ensure potential inhibition. 24 hours plasma samples were withdrawn, area under the curve (AUC) ratios were calculated and compared to the basal state. After an end of study visit on the day of the 24h blood sample (following the second study day), probands were discharged.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged between 18 and 45 years (inclusive) at screening
* BMI between 18 and 28 kg/m2 (inclusive) and bodyweight at least 50 kg at screening
* systolic blood pressure: 100-140 mmHg, diastolic blood pressure: 60-90 mmHg and heart rate: 45-90 bpm (inclusive), measured on the leading arm, in the supine position at screening
* No clinically significant findings on the physical examination at screening
* Signed informed consent prior to any study-mandated procedure
* Hematology and clinical chemistry results not deviating from the normal range to clinically relevant extent at screening
* Ability to communicate well with the investigator to understand and comply with the requirements of the study

Exclusion Criteria:

* Smoking >5 cigarettes per day
* History or clinical evidence of alcoholism or drug abuse within the 3- year period prior to screening
* Loss of ≥250 ml of blood within 3 months prior to screening. Treatment with an investigational drug within 30 days prior to screening
* Previous systemic treatment with any prescribed or over the counter medication (including herbal medicines such as St John's Wort) within 2 weeks prior to the intended start of the study
* Inability to stop consumption inducing food products (e.g. grapefruit juice) 72 h before start of the study
* Excessive caffeine consumption (>8 cups of coffee/ 8l coca cola per day)
* Legal incapacity or limited legal capacity at screening
* Positive results from urine drug screen at screening
* History or clinical evidence of any disease (e.g. gastrointestinal disease: Morbus Crohn, Colitis Ulcerosa, anamnestic gastrointestinal bleeding) and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drugs, or which might increase the risk for toxicity
* Known hypersensitivity to Metamizole (Novalgin®) or excipients of the drug formulation
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Effect on AUC ratio between parent and metabolite | 12 hours
  AUC ratio between parent and metabolite of specific cytochrome P450 substrates to determine a shift which may indicate either induction or inhibition of the specific cytochrome P450
Cmax | 24 hours
  Maximal Concentration in plasma of parent and metabolite
tmax | 24 hours
  time to reach Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Krähenbühl, Prof. Dr. MD, Principal Investigator — Head of Clinical Pharmacology, University Hospital Basel
Locations (1):
- Clinical Trial Unit, University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No